CLINICAL TRIAL: NCT05356338
Title: Expanding Reach of a Health System Intervention for Family Beverage Choice by Partnering With a Local WIC Program
Brief Title: Expanding Health System Intervention Through The Women, Infants and Children (WIC) Program Partnership
Acronym: WHISPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00073800
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-04

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff collecting data on the primary outcome of beverage consumption at 3 and 6 month follow-up will be blinded to group allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group participants in this study will not receive any intervention as is the current standard of clinical care for excess sugary drink consumption. They will receive monthly check-in reminders from research staff to promote engagement and retention and will participate in data collection visits at baseline, 3 and 6 months.
- Intervention (Experimental): Intervention participants will receive a 6-month behavioral intervention with the following components: A water promotion toolkit that includes water bottles, water flavor infusers, stickers to decorate bottles, children's book about water consumption, and instructions for other intervention components (how to view videos, download app, and prepare for calls) Two brief educational videos: a 5-minute video about healthy drink choices for the family and a 3-min video educating residents about local water. Ready, Set Gulp! app for families that will help all family members track their beverage intake, find out how much water and sugar they are consuming, set goals, compete for points, answer quiz questions and create new recipes for flavor infused water. A series of 14 interactive voice response phone calls to parents over 6 months that educate parents on topics relevant to improving family drink choices.
  Two counseling sessions by a WIC nutritionist at months 2 and 4
  Interventions: Behavioral: Pilot Intervention to reduce SSB consumption in children and families enrolled in WIC

INTERVENTIONS:
Behavioral: Pilot Intervention to reduce SSB consumption in children and families enrolled in WIC — A 6-month intervention based on the use of 5 components: 2 educational videos, provision of a water-promotion "toolkit," a mobile phone application (app), a series of 14 computerized interactive voice response (IVR) phone calls to parents and 2 counseling sessions by a WIC nutritionist to compare families' SSB's consumption behaviors
  Arms: Intervention

SUMMARY:
Pilot test the health system-based intervention to improve family beverage choices and promote water consumption, engaging WIC nutritionists to augment the intervention with follow-up and counseling of families at regularly-scheduled WIC appointments in a small randomized trial among 30 WIC-enrolled families.

DETAILED DESCRIPTION:
This is a pilot 2-arm randomized trial among 30 WIC enrolled families of children 6 months through 4 years old who currently over-consume sugary drinks. The study team will randomize families to either an intervention group, that will receive a behavioral intervention consisting of two educational videos, a water promotion toolkit, mobile phone app, series of educational phone calls and extra counseling from WIC nutritionists, or to a control group that will not receive this intervention. The study team will compare 6-month change in child and parental beverage consumption between groups. Exploratory analyses will examine child weight (kg) and Body Mass Index (BMI) z-score (BMIz) outcomes, and compare intervention effects across race/ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Child 6 months - 4 years old who receives health care attention at Wake Forest pediatric or family medicine practices
* Child enrolled in WIC
* Child consumes 2 or more SSB and/or fruit juice total per day
* Child with no chronic health condition
* Child has not seen nutritionist or visited our family-based weight management clinic in the past year
* Parent/caregiver who has not watch educational video "Get in the Zero Zone"
* Parent/caregiver has a smartphone and reliable internet
* Parent/caregiver able to communicate well in English

Exclusion Criteria:

* Child doesn't meet age criteria
* Child consumes less than 2 SSB and/or fruit juice total per day
* Child with a chronic health condition
* Child has seen nutritionist or visited our family-based weight management clinic in the past year
* Parent/caregiver has watched educational video "Get in the Zero Zone"
* Parent/caregiver has completed interview or usability test
* Parent/caregiver doesn't have a smartphone or reliable internet
* Parent/caregiver not able to communicate well in English

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change in child sugary drink serving consumption | from baseline to month 3
  change in a child's combined consumption of Sugar-Sweetened Beverages (SSB)+Fruit Juice (FJ), measured as total servings per day, at 3 and 6 months after starting intervention, measured with Beverage Intake Questionnaire (BevQ15) instrument
Change in child sugary drink serving consumption | from baseline to month 6
  change in a child's combined consumption of Sugar-Sweetened Beverages (SSB)+Fruit Juice (FJ), measured as total servings per day, at 3 and 6 months after starting intervention, measured with Beverage Intake Questionnaire (BevQ15) instrument

SECONDARY OUTCOMES:
BevQ 15 - Children Change in Servings of Water Consumption | from baseline to month 3, from baseline to month 6
  changes in total servings of water consumed by children
BevQ 15 - Children Change in Servings of SSBs Consumption | from baseline to month 3, from baseline to month 6
  changes in total servings of SSBs consumed by children
BevQ 15 - Children Change in Servings of 100% Fruit Juice Consumption | from baseline to month 3, from baseline to month 6
  changes in total servings of 100% fruit juice consumed by children
BevQ 15 - Children Change in total Volume of Water Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume of water consumed by children
BevQ 15 - Children Change in total Volume of SSBs Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume of SSBs consumed by children
BevQ 15 - Children Change in total Volume of 100% Fruit Juice Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume of 100% fruit juice consumed by children
BevQ 15 - Children Change in total calories of beverages consumption | from baseline to month 3, from baseline to month 6
  Changes in calories of beverages consumed by children
BevQ 15 -Parental Change in Servings of Water Consumption | from baseline to month 3, from baseline to month 6
  Changes in total servings of water consumed by parents
BevQ 15 -Parental Change in Servings of SSBs Consumption | from baseline to month 3, from baseline to month 6
  Changes in total servings of SSBs consumed by parents
BevQ 15 -Parental Change in Servings of 100% Fruit Juice Consumption | from baseline to month 3, from baseline to month 6
  Changes in total servings of 100% fruit juice consumed by parents
BevQ 15 -Parental Change in Volume of Water Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume of water consumed by parents
BevQ 15 -Parental Change in Volume of SSBs Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume of SSBs consumed by parents
BevQ 15 -Parental Change in Volume of 100% fruit juice Consumption | from baseline to month 3, from baseline to month 6
  changes in total volume of 100% fruit juice consumed by parents
BevQ 15-Parental Change in Calories of Beverage Consumption | from baseline to month 3, from baseline to month 6
  changes in total beverage calories for parents
Changes in parent knowledge | from baseline, month 6
  Survey knowledge items will be "scored" in terms of correct or not with a range of 0-17 possible points, with higher score demonstrating more knowledge about SSB and FJ.
Changes in Parent Attitudes | from baseline, month 6
  Attitude and belief items will be reported individually, as these are not objectively correct or incorrect and represent a subjective state of the parent's point of view. These will be reported out as frequencies / descriptive statistics, with change in proportion responding a certain way examined over follow-up. Statistician will use Statistical Analysis Software (SAS) for quantifying qualitative data.
Changes in Parent Beliefs | from baseline, month 6
  Belief items will be reported individually, as these are not objectively correct or incorrect and represent a subjective state of the parent's point of view. These will be reported out as frequencies / descriptive statistics, with change in proportion responding a certain way examined over follow-up. Statistician will use Statistical Analysis Software (SAS) for quantifying qualitative data.
Child Weight Change | from baseline to month 3, from baseline to month 6
  change in child weight (kg) using Electronic Health Record (EHR) data
Child Body Mass Index Z-Score (BMIz) Change | from baseline to month 3, from baseline to month 6
  change in child BMIz also using EHR data

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Lewis, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT05356338/ICF_000.pdf